CLINICAL TRIAL: NCT06899620
Title: Weizmannia Coagulans BC179 Alleviates Post-Alcohol Discomfort May Via Taurine-Related Metabolism and Antioxidant Regulation: A Randomized, Double-Blind，Placebo-Controlled Trial
Brief Title: BC179 Relieves Discomfort After Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: WK20250323
Record Dates: First submitted 2025-03-25; First posted 2025-03-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Drinking Behavior
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 10B CFU/Sachet/Day BC179 ; Storage: Store in cool and dry place without sun exposure
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): Dextrin one Sachet/Day; Storage: Store in cool and dry place without sun exposure
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — The experimental phase of this study lasted for 60 days.
  Arms: Probiotic group
Dietary Supplement: Placebo group — The experimental phase of this study lasted for 60 days.
  Arms: Placebo group

SUMMARY:
To assess the effectiveness and safety of probiotic strain BC179 in reducing alcohol absorption in the gut, thereby lowering health risks.

ELIGIBILITY:
* Inclusion Criteria:

  1. Participants must be aged between 18 and 65 years.
  2. They should have a documented history of long-term alcohol consumption, defined as consuming at least 20 grams of ethanol per day for at least one year. This is calculated using the formula: volume (mL) × alcohol content (%) × 0.8.
  3. They must provide written informed consent and be willing to comply with the study procedures.
* Exclusion Criteria:

  1. History of chronic liver, gastrointestinal, or systemic metabolic disorders.
  2. Use of products with similar functions to the investigational formulation within the past two weeks.
  3. Use of antibiotics, laxatives, or dietary supplements within the past four weeks.
  4. Documented history of hypertension or diabetes.
  5. Severe allergies or immune deficiencies.
  6. Pregnancy, lactation, or planning pregnancy without effective contraception during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Effects of BC179 on alcohol metabolism | 60 days
  The impact of BC179 on alcohol metabolism is assessed by monitoring blood alcohol concentration (BAC) and related enzyme activities, such as alcohol dehydrogenase (ADH) and aldehyde dehydrogenase (ALDH).

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Ying, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No